CLINICAL TRIAL: NCT04292977
Title: Splanchnic and Systemic VLDL-TG and FFA Balance in Individuals With NAFL and NASH
Brief Title: Splanchnic and Systemic VLDL-TG and FFA Balance
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Other Study IDs: Jeyanthini
Record Dates: First submitted 2020-02-28; First posted 2020-03-03 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2022-05

CONDITIONS: NAFLD; NASH - Nonalcoholic Steatohepatitis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To determine differences between NAFLD and NASH subjects with respect to hepatic FA metabolism (uptake, oxidation, and re-esterification) and hepatic VLDL-TG secretion and peripheral kinetics (oxidation and tissue storage). 8 non-diabetic upper-body obese subjects with NAFLD and 8 with NASH (biopsy proven) will be studied in the overnight fasted state. VLDL-TG stable isotope will be used in combination with hepatic vein catherization to directly measure splanchnic VLDL-TG uptake and secretion. FFA (palmitate) tracers as well as adipose tissue and skeletal muscle biopsies will be used to measure whole-body substrate turnover and flexibility as well as tissue specific substrate handling during fasting and hyperinsulinemic conditions.

ELIGIBILITY:
Inclusion Criteria:

* 8 obese subject men with NAFL (MR spectroskopi, fibro scanner) (BMI > 28).
* 8 obese subject men with NASH (MR spectroskopi, fibro scanner) (BMI > 28). age between 40-70 years. Written consent before the start of the study.

Exclusion Criteria:

* known current disease
* fixed medical drug consumption except antihypertensive drugs and statins. However, pause statins 3 weeks before the examination date Blood donation within the last 3 months prior to the study Participation in experiments involving radioactive isotopes within the last 3 months Alcohol abuse (over 21 items per week for men and 14 for women) Smoking Weight over 130 kg Cancer patients Large intake of medication

Ages: 40 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 8 obese subject men with NAFL (MR spectroskopi, fibro scanner) (BMI > 28).
  - 8 obese subject men with NASH (MR spectroskopi, fibro scanner) (BMI > 28). age between 40-70 years.
Sampling Method: Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2020-11-15 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
Splanchnic and systemic VLDL-TG and FFA balance in individuals with biopsy proven NAFL or NASH | 2 years
  splanchnic (liver) VLDL-TG and FFA uptake and secretion, in individuals with biopsy proven NAFL or NASH

CONTACTS AND LOCATIONS:
Locations (1):
- Arhus University Hospital Department of Endocrinology and Internal Medicine Skejby, Aarhus N, Denmark, 8200, Skejby, Aarhus N, Denmark

REFERENCES:
- [Derived] Risikesan J, Heeboll S, Kumarathas I, Sondergaard E, Johansen RF, Ringgaard S, Aagaard NK, Sandahl TD, Villadsen GE, Gormsen LC, Frystyk J, Jensen MD, Gronbaek H, Nielsen S. Similar insulin regulation of splanchnic FFA and VLDL-TG in men with nonalcoholic hepatic steatosis and steatohepatitis. J Lipid Res. 2024 Jul;65(7):100580. doi: 10.1016/j.jlr.2024.100580. Epub 2024 Jun 18. PMID 38901559